CLINICAL TRIAL: NCT00481767
Title: Study to Assess the Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' HPV Vaccine GSK580299 in Healthy Female Subjects Aged 10-25 Years.
Brief Title: Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) Vaccine (GSK580299) in Healthy Female Subjects 10-25 Years of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 106069; 2017-000416-42 (EudraCT Number)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Human Papillomavirus (HPV) Infection
Keywords: Safety; Immunogenicity; Human Papillomavirus (HPV) vaccine
MeSH Terms: conditions — Papillomavirus Infections; Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervarix Group (Active Comparator): Healthy female subjects who received 3 doses of Cervarix at Months 0, 1 and 6, administered intramuscularly into the deltoid region of the non-dominant arm. For some analyses the group was stratified by age into a 10-14 years of age group and a 15-25 years of age group.
  Interventions: Biological: Cervarix
- Placebo Group (Placebo Comparator): Healthy female subjects who received 3 doses of placebo at Months 0, 1 and 6, administered intramuscularly into the deltoid region of the non-dominant arm. For some analyses the group was stratified by age into a 10-14 years of age group and a 15-25 years of age group.
  Interventions: Drug: Placebo Al(OH)3

INTERVENTIONS:
Biological: Cervarix — The vaccine was administered according to a 0, 1, and 6-month schedule, intramuscularly into the deltoid region of the non-dominant arm.
  Other Names: GlaxoSmithKline Biologicals' HPV vaccine GSK580299; HPV-16/18 L1 AS04 vaccine
  Arms: Cervarix Group
Drug: Placebo Al(OH)3 — Placebo was administered according to a 0, 1 and 6-month schedule, intramuscularly into the deltoid region of the non-dominant arm.
  Arms: Placebo Group

SUMMARY:
Cervical cancer is the second most common cancer among women worldwide. Approximately 500 000 new cases are reported each year worldwide, from which 83% occur in developing countries. The incidence of cervical cancer varies depending on the region of the world. Africa has some of the highest age-standardized incidence and mortality rates in the world (Eastern Africa 42.7 and 34.6 per 100 000; Southern Africa 38.2 and 22.6 per 100 000; Western Africa 29.3 and 23.8 per 100 000; Middle Africa 28.0 and 23.0 per 100 000).

As in the majority of developing countries, organization of cervical cancer screening programs in Africa is difficult to manage, especially in rural areas. HPV prophylactic vaccination could therefore clearly and efficiently decrease the incidence of cervical cancer. The current study is designed to assess the immunogenicity and safety of GSK Biologicals' HPV-16/18 L1 AS04 vaccine in female subjects enrolled from multiple countries in Africa.

Ideally, HPV vaccination should be performed before onset of sexual activity, since studies have shown that acquisition of high-risk HPV occurs soon after sexual debut. This study will therefore be performed in subjects aged 10 to 25 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents/legally acceptable representative can and will comply with the requirements of the protocol should be enrolled in the study.
* A female between, and including, 10 and 25 years of age at the time of the first vaccination.
* Written or oral, signed or thumb printed or witnessed informed consent obtained from the subject prior to enrolment. For subjects below legal age of consent, written or oral, signed or thumb printed or witnessed informed consent obtained from the subject's parent or legally acceptable representative. In addition, a written or oral, signed or thumb printed and witnessed informed assent must be obtained from the subject.
* Free of obvious health problems as established by medical history, clinical examination and laboratory testing before entering into the study.
* Subjects must have a negative urine pregnancy test at the screening visit and at Visit 1 (Day 0).
* Subjects must be seronegative for human immunodeficiency virus (HIV) at the screening visit.
* Subjects must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series. Subjects who reach menarche during the study and therefore are of childbearing potential must agree to follow the same precautions.
* Subjects must have had no more than 6 sexual partners prior to enrolment.
* Subjects must be willing to undergo HIV voluntary counselling and testing and must be willing to be informed of their HIV status. Subjects below legal age of consent must also be willing to have their parent or legally acceptable representative informed of their HIV status.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 12).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine. Enrolment will be deferred until the subject is outside of specified window.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after any dose of study vaccine.
* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Previous administration of components of the investigational vaccine.
* Cancer or autoimmune disease under treatment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection based on laboratory testing performed during the screening visit.
* Hypersensitivity to latex.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine/control.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory testing performed at the screening visit.
* History of any neurologic disorders or seizures.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or breastfeeding female.
* A women planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period, up to two months after the last vaccine dose.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 676 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2010-02-25 (Actual); Study Completion 2010-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Dakar, Senegal
- GSK Investigational Site, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kiviat N et al. Immunisation of African pre-teen/adolescent girls and young women with the HPV-16/18 AS04-adjuvanted vaccine. Abstract presented at South African Society of Obstetricians and Gynaecologists - O & G Update 2011. Pretoria, South Africa, 5-7 May 2011.
- [Background] Sow PS, Watson-Jones D, Kiviat N, Changalucha J, Mbaye KD, Brown J, Bousso K, Kavishe B, Andreasen A, Toure M, Kapiga S, Mayaud P, Hayes R, Lebacq M, Herazeh M, Thomas F, Descamps D. Safety and immunogenicity of human papillomavirus-16/18 AS04-adjuvanted vaccine: a randomized trial in 10-25-year-old HIV-Seronegative African girls and young women. J Infect Dis. 2013 Jun 1;207(11):1753-63. doi: 10.1093/infdis/jis619. Epub 2012 Dec 13. PMID 23242542
- [Background] Sow PS. et al. Immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine in African preteen/adolescent girls and young women. Abstract presented at the African Organisation for Research and Training in Cancer (AORTIC). Cairo, Egypt, November 30 - December 3, 2011.
- [Background] Watson-Jones D, Baisley K, Brown J, Kavishe B, Andreasen A, Changalucha J, Mayaud P, Kapiga S, Gumodoka B, Hayes RJ, de Sanjose S. High prevalence and incidence of human papillomavirus in a cohort of healthy young African female subjects. Sex Transm Infect. 2013 Aug;89(5):358-65. doi: 10.1136/sextrans-2012-050685. Epub 2013 Mar 13. PMID 23486859
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 106069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix Group | Placebo Group
Started | 450 | 226
Completed | 418 | 205
Not Completed | 32 | 21
Not completed — Withdrawal by Subject | 16 | 11
Not completed — Lost to Follow-up | 16 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Placebo Group | Total
Number analyzed (Participants) | 450 | 226 | 676
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.9 (4.36) | 16.8 (4.16) | 16.9 (4.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 450 | 226 | 676
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/African american | 431 | 219 | 650
  Not specified | 19 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti-human Papillomavirus (HPV)-16 and 18 Antibodies
Description: A seroconverted subject was a subject with antibody titers below 8 or 7 Enzyme-linked Immunosorbent Assay Units per milliliter (EL.U/mL) for anti-HPV-16 and 18, respectively, before vaccination and antibody titers ≥ 8 or 7 EL.U/mL for anti-HPV-16 and 18, respectively, after vaccination. The groups were stratified by age for the analysis. The age strata were 10-14 years and 15-25 years.
Time Frame: At Month 7
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 212 | 98
Participants
  10-14 years anti-HPV-16: number analyzed (Participants) | 130 | 59
  10-14 years anti-HPV-16 | 130 | 4
  15-25 years anti-HPV-16: number analyzed (Participants) | 190 | 97
  15-25 years anti-HPV-16 | 190 | 5
  10-14 years anti-HPV-18: number analyzed (Participants) | 128 | 56
  10-14 years anti-HPV-18 | 128 | 2
  15-25 years anti-HPV-18 | 212 | 5

2. Primary Outcome: Geometric Mean Titers (GMTs) of Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: Titers were expressed as GMTs in Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL). The groups were stratified by age for the analysis. The age strata were 10-14 years and 15-25 years.
Time Frame: At Month 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 237 | 114
EL.U/mL
  10-14 years anti-HPV-16: number analyzed (Participants) | 142 | 65
  10-14 years anti-HPV-16 | 18591.3 [16433.0 to 21033.1] | 4.8 [4.2 to 5.5]
  15-25 years anti-HPV-16: number analyzed (Participants) | 237 | 112
  15-25 years anti-HPV-16 | 10664.0 [9668.5 to 11762.0] | 5.3 [4.6 to 6.1]
  10-14 years anti-HPV-18: number analyzed (Participants) | 141 | 66
  10-14 years anti-HPV-18 | 6409.8 [5563.4 to 7385.0] | 3.9 [3.6 to 4.2]
  15-25 years anti-HPV-18: number analyzed (Participants) | 235 | 114
  15-25 years anti-HPV-18 | 3653.6 [3343.9 to 3991.9] | 4.6 [4.0 to 5.3]

3. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: as for outcome 1
Time Frame: At Month 2 and Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 212 | 98
Participants
  10-14 years anti-HPV-16 Month 2: number analyzed (Participants) | 130 | 59
  10-14 years anti-HPV-16 Month 2 | 130 | 1
  15-25 years anti-HPV-16 Month 2: number analyzed (Participants) | 190 | 96
  15-25 years anti-HPV-16 Month 2 | 190 | 3
  10-14 years anti-HPV-16 Month 12: number analyzed (Participants) | 128 | 59
  10-14 years anti-HPV-16 Month 12 | 128 | 2
  15-25 years anti-HPV-16 Month 12: number analyzed (Participants) | 184 | 94
  15-25 years anti-HPV-16 Month 12 | 184 | 7
  10-14 years anti-HPV-18 Month 2: number analyzed (Participants) | 128 | 55
  10-14 years anti-HPV-18 Month 2 | 128 | 1
  15-25 years anti-HPV-18 Month 2 | 212 | 4
  10-14 years anti-HPV-18 Month 12: number analyzed (Participants) | 126 | 56
  10-14 years anti-HPV-18 Month 12 | 125 | 0
  15-25 years anti-HPV-18 Month 12: number analyzed (Participants) | 205 | 96
  15-25 years anti-HPV-18 Month 12 | 205 | 6

4. Secondary Outcome: GMTs for Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: as for outcome 2
Time Frame: At Month 2 and Month 12
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 237 | 112
EL.U/mL
  10-14 years anti-HPV-16 Month 2: number analyzed (Participants) | 142 | 64
  10-14 years anti-HPV-16 Month 2 | 5340.2 [4823.7 to 5912.0] | 4.5 [4.0 to 5.0]
  15-25 years anti-HPV-16 Month 2 | 3732.6 [3436.6 to 4054.1] | 4.9 [4.3 to 5.5]
  10-14 years anti-HPV-16 Month 12: number analyzed (Participants) | 139 | 65
  10-14 years anti-HPV-16 Month 12 | 4016.2 [3323.3 to 4853.7] | 4.7 [4.2 to 5.3]
  15-25 years anti-HPV-16 Month 12: number analyzed (Participants) | 229 | 109
  15-25 years anti-HPV-16 Month 12 | 2464.2 [2196.5 to 2764.5] | 5.6 [4.7 to 6.6]
  10-14 years anti-HPV-18 Month 2: number analyzed (Participants) | 141 | 65
  10-14 years anti-HPV-18 Month 2 | 3016.7 [2677.4 to 3398.9] | 3.9 [3.6 to 4.3]
  15-25 years anti-HPV-18 Month 2: number analyzed (Participants) | 235 | 112
  15-25 years anti-HPV-18 Month 2 | 2039.3 [1861.3 to 2234.4] | 4.6 [4.0 to 5.3]
  10-14 years anti-HPV-18 Month 12: number analyzed (Participants) | 138 | 66
  10-14 years anti-HPV-18 Month 12 | 1422.1 [1170.0 to 1728.4] | 3.7 [3.5 to 3.9]
  15-25 years anti-HPV-18 Month 12: number analyzed (Participants) | 227 | 111
  15-25 years anti-HPV-18 Month 12 | 855.9 [768.3 to 953.5] | 4.6 [4.0 to 5.4]

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain and swelling at the injection site. Any = occurrence of any solicited local symptom regardless of their intensity grade. Grade 3 swelling = swelling spreading beyond 50 millimeters (mm) of injection site. Grade 3 pain = pain that prevented normal activity.
Time Frame: Within 7 days (Day 0-6) after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 450 | 226
Participants
  Any Pain, Dose 1 | 309 | 116
  Grade 3 Pain, Dose 1 | 2 | 0
  Any Swelling, Dose 1 | 15 | 7
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 437 | 217
  Any Pain, Dose 2 | 265 | 95
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Pain, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 437 | 217
  Any Swelling, Dose 2 | 45 | 15
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 411 | 200
  Any Pain, Dose 3 | 200 | 66
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Pain, Dose 3 | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 411 | 200
  Any Swelling, Dose 3 | 26 | 10
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Swelling, Dose 3 | 0 | 0
  Any Pain, Across doses | 375 | 166
  Grade 3 Pain, Across doses | 2 | 0
  Any Swelling, Across doses | 74 | 27
  Grade 3 Swelling, Across doses | 0 | 0

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia (only joints that are distal from the injection site), fatigue, fever (defined as axillary temperature ≥ 37.5 degrees Celsius), gastrointestinal symptoms, headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 urticaria = urticaria distributed on at least 4 body areas. Grade 3 fever = axillary temperature > 39.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 7 days (Day 0-6) after each dose and across doses
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 450 | 226
Participants
  Any Arthralgia, Dose 1 | 19 | 10
  Grade 3 Arthralgia, Dose 1 | 0 | 0
  Related Arthralgia, Dose 1 | 7 | 2
  Any Fatigue, Dose 1 | 34 | 12
  Grade 3 Fatigue, Dose 1 | 0 | 0
  Related Fatigue, Dose 1 | 21 | 3
  Any Fever, Dose 1 | 72 | 43
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 34 | 17
  Any Gastrointestinal, Dose 1 | 34 | 21
  Grade 3 Gastrointestinal, Dose 1 | 0 | 0
  Related Gastrointestinal, Dose 1 | 14 | 8
  Any Headache, Dose 1 | 89 | 56
  Grade 3 Headache, Dose 1 | 0 | 0
  Related Headache, Dose 1 | 51 | 25
  Any Myalgia, Dose 1 | 35 | 16
  Grade 3 Myalgia, Dose 1 | 0 | 0
  Related Myalgia, Dose 1 | 22 | 7
  Any Rash, Dose 1 | 14 | 8
  Grade 3 Rash, Dose 1 | 0 | 0
  Related Rash, Dose 1 | 1 | 0
  Any Urticaria, Dose 1 | 12 | 7
  Grade 3 Urticaria, Dose 1 | 0 | 0
  Related Urticaria, Dose 1 | 0 | 0
  Any Arthralgia, Dose 2: number analyzed (Participants) | 437 | 217
  Any Arthralgia, Dose 2 | 47 | 17
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Arthralgia, Dose 2 | 0 | 0
  Related Arthralgia, Dose 2: number analyzed (Participants) | 437 | 217
  Related Arthralgia, Dose 2 | 4 | 2
  Any Fatigue, Dose 2: number analyzed (Participants) | 437 | 217
  Any Fatigue, Dose 2 | 62 | 25
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Fatigue, Dose 2 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 437 | 217
  Related Fatigue, Dose 2 | 17 | 4
  Any Fever, Dose 2: number analyzed (Participants) | 437 | 217
  Any Fever, Dose 2 | 82 | 33
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 437 | 217
  Related Fever, Dose 2 | 19 | 8
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 437 | 217
  Any Gastrointestinal, Dose 2 | 66 | 26
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 437 | 217
  Related Gastrointestinal, Dose 2 | 15 | 6
  Any Headache, Dose 2: number analyzed (Participants) | 437 | 217
  Any Headache, Dose 2 | 96 | 49
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Headache, Dose 2 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 437 | 217
  Related Headache, Dose 2 | 40 | 18
  Any Myalgia, Dose 2: number analyzed (Participants) | 437 | 217
  Any Myalgia, Dose 2 | 50 | 17
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Myalgia, Dose 2 | 0 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 437 | 217
  Related Myalgia, Dose 2 | 9 | 3
  Any Rash, Dose 2: number analyzed (Participants) | 437 | 217
  Any Rash, Dose 2 | 44 | 15
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Rash, Dose 2 | 0 | 0
  Related Rash, Dose 2: number analyzed (Participants) | 437 | 217
  Related Rash, Dose 2 | 1 | 0
  Any Urticaria, Dose 2: number analyzed (Participants) | 437 | 217
  Any Urticaria, Dose 2 | 43 | 14
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 437 | 217
  Grade 3 Urticaria, Dose 2 | 0 | 0
  Related Urticaria, Dose 2: number analyzed (Participants) | 437 | 217
  Related Urticaria, Dose 2 | 0 | 0
  Any Arthralgia, Dose 3: number analyzed (Participants) | 411 | 200
  Any Arthralgia, Dose 3 | 28 | 10
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Arthralgia, Dose 3 | 0 | 0
  Related Arthralgia, Dose 3: number analyzed (Participants) | 411 | 200
  Related Arthralgia, Dose 3 | 0 | 0
  Any Fatigue, Dose 3: number analyzed (Participants) | 411 | 200
  Any Fatigue, Dose 3 | 34 | 13
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Fatigue, Dose 3 | 0 | 0
  Related Fatigue, Dose 3: number analyzed (Participants) | 411 | 200
  Related Fatigue, Dose 3 | 4 | 3
  Any Fever, Dose 3: number analyzed (Participants) | 411 | 200
  Any Fever, Dose 3 | 81 | 33
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Fever, Dose 3 | 0 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 411 | 200
  Related Fever, Dose 3 | 20 | 9
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 411 | 200
  Any Gastrointestinal, Dose 3 | 43 | 19
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Gastrointestinal, Dose 3 | 0 | 0
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 411 | 200
  Related Gastrointestinal, Dose 3 | 5 | 5
  Any Headache, Dose 3: number analyzed (Participants) | 411 | 200
  Any Headache, Dose 3 | 71 | 33
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Headache, Dose 3 | 0 | 0
  Related Headache, Dose 3: number analyzed (Participants) | 411 | 200
  Related Headache, Dose 3 | 22 | 12
  Any Myalgia, Dose 3: number analyzed (Participants) | 411 | 200
  Any Myalgia, Dose 3 | 28 | 10
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Myalgia, Dose 3 | 0 | 0
  Related Myalgia, Dose 3: number analyzed (Participants) | 411 | 200
  Related Myalgia, Dose 3 | 1 | 0
  Any Rash, Dose 3: number analyzed (Participants) | 411 | 200
  Any Rash, Dose 3 | 26 | 12
  Grade 3 Rash, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Rash, Dose 3 | 0 | 0
  Related Rash, Dose 3: number analyzed (Participants) | 411 | 200
  Related Rash, Dose 3 | 0 | 0
  Any Urticaria, Dose 3: number analyzed (Participants) | 411 | 200
  Any Urticaria, Dose 3 | 26 | 11
  Grade 3 Urticaria, Dose 3: number analyzed (Participants) | 411 | 200
  Grade 3 Urticaria, Dose 3 | 0 | 0
  Related Urticaria, Dose 3: number analyzed (Participants) | 411 | 200
  Related Urticaria, Dose 3 | 0 | 0
  Any Arthralgia, Across doses | 77 | 32
  Grade 3 Arthralgia, Across doses | 0 | 0
  Related Arthralgia, Across doses | 10 | 4
  Any Fatigue, Across doses | 111 | 42
  Grade 3 Fatigue, Across doses | 0 | 0
  Related Fatigue, Across doses | 39 | 9
  Any Fever, Across doses | 147 | 70
  Grade 3 Fever, Across doses | 0 | 0
  Related Fever, Across doses | 57 | 27
  Any Gastrointestinal, Across doses | 118 | 56
  Grade 3 Gastrointestinal, Across doses | 0 | 0
  Related Gastrointestinal, Across doses | 31 | 17
  Any Headache, Across doses | 189 | 109
  Grade 3 Headache, Across doses | 0 | 0
  Related Headache, Across doses | 101 | 46
  Any Myalgia, Across doses | 90 | 36
  Grade 3 Myalgia, Across doses | 0 | 0
  Related Myalgia, Across doses | 27 | 9
  Any Rash, Across doses | 71 | 30
  Grade 3 Rash, Across doses | 0 | 0
  Related Rash, Across doses | 2 | 0
  Any Urticaria, Across doses | 68 | 27
  Grade 3 Urticaria, Across doses | 0 | 0
  Related Urticaria, Across doses | 0 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity and relationship to vaccination. Grade 3 = an unsolicited AE that prevented normal everyday activity. Related = unsolicited AE assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 30 days (Day 0-29) after any vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 450 | 226
Participants
  Any AE(s) | 235 | 142
  Grade 3 AE(s) | 5 | 1
  Related AE(s) | 3 | 4

8. Secondary Outcome: Number of Subjects With NOCDs and Other MSCs
Description: New onset of chronic diseases (NOCDs) assessed included autoimmune disorders, asthma, type I diabetes, allergies. Medically significant conditions (MSCs) assessed included AEs prompting emergency room or physician visits that were not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that were not related to common diseases. Common diseases included upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 up to Month 7 and from Month 7 up to Month 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 450 | 226
Participants
  NOCD(s) up to Month 7 | 10 | 8
  NOCD(s) Month 7-12: number analyzed (Participants) | 421 | 208
  NOCD(s) Month 7-12 | 1 | 3
  MSC(s) up to Month 7 | 289 | 161
  MSC(s) Month 7-12: number analyzed (Participants) | 421 | 208
  MSC(s) Month 7-12 | 121 | 68

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 7 and from Month 7 up to Month 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 450 | 226
Participants
  up to Month 7 | 12 | 10
  up to Month 12 | 17 | 14

10. Secondary Outcome: Number of Subjects With Pregnancies and Their Outcomes
Description: Pregnancy outcomes were ectopic pregnancy, elective termination no apparent congenital anomaly, live infant no apparent congenital anomaly, premature live infant no apparent congenital anomaly, lost to follow-up and spontaneous abortion no apparent congenital anomaly.
Time Frame: From Day 0 up to Month 12
Population: The analysis was performed on the Total Vaccinated cohort, which included vaccinated subjects with at least one vaccine administration documented and who reported pregnancies (and their outcomes).
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 14 | 10
Participants
  Ectopic pregnancy | 1 | 0
  Elective termination | 3 | 3
  Live infant | 5 | 5
  Premature live infant | 3 | 1
  Lost to follow-up | 1 | 0
  Spontaneous abortion | 1 | 1

11. Secondary Outcome: Number of Senegalese Subjects With Clinically Relevant Abnormalities in Parameters Assessed
Description: Biochemical and haematological parameters assessed were: Alanine amino-transferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), hematocrit (HC), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), white blood cells (WBC). Number of subjects were separated with respect to their results at pre-vaccination, i.e. whether their results were in, above or below the normal range. N for each category at pre-vaccination noted in category title. For each parameter and for each range it was assessed whether the values of the subjects were in, above or below the normal range.
Time Frame: At Month 7
Population: The analysis was performed on the Total Vaccinated cohort on Senegalese subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 217 | 105
Participants
  ALT, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 8 | 4
  ALT, pre-vacc. ABOVE, Month 7 NORMAL | 7 | 4
  ALT, pre-vacc.ABOVE, Month 7 BELOW: number analyzed (Participants) | 8 | 4
  ALT, pre-vacc.ABOVE, Month 7 BELOW | 0 | 0
  ALT, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 8 | 4
  ALT, pre-vacc. ABOVE, Month 7 ABOVE | 1 | 0
  ALT, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 39 | 17
  ALT, pre-vacc. BELOW, Month 7 NORMAL | 15 | 7
  ALT, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 39 | 17
  ALT, pre-vacc. BELOW, Month 7 BELOW | 24 | 10
  ALT, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 39 | 17
  ALT, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  ALT, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 170 | 84
  ALT, pre-vacc. NORMAL, Month 7 NORMAL | 137 | 57
  ALT, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 170 | 84
  ALT, pre-vacc. NORMAL, Month 7 BELOW | 30 | 25
  ALT, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 170 | 84
  ALT, pre-vacc. NORMAL, Month 7 ABOVE | 3 | 2
  BAS, pre-vacc. NORMAL, Month 7 NORMAL | 216 | 105
  BAS, pre-vacc. NORMAL, Month 7 BELOW | 0 | 0
  BAS, pre-vacc. NORMAL, Month 7 ABOVE | 1 | 0
  CREA, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 2 | 1
  CREA, pre-vacc. ABOVE, Month 7 NORMAL | 1 | 1
  CREA, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 2 | 1
  CREA, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  CREA, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 2 | 1
  CREA, pre-vacc. ABOVE, Month 7 ABOVE | 1 | 0
  CREA, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 56 | 30
  CREA, pre-vacc. BELOW, Month 7 NORMAL | 19 | 13
  CREA, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 56 | 30
  CREA, pre-vacc. BELOW, Month 7 BELOW | 37 | 17
  CREA, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 56 | 30
  CREA, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  CREA, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 159 | 74
  CREA, pre-vacc. NORMAL, Month 7 NORMAL | 149 | 68
  CREA, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 159 | 74
  CREA, pre-vacc. NORMAL, Month 7 BELOW | 10 | 4
  CREA, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 159 | 74
  CREA, pre-vacc. NORMAL, Month 7 ABOVE | 0 | 2
  EOS, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 43 | 28
  EOS, pre-vacc. ABOVE, Month 7 NORMAL | 9 | 12
  EOS, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 43 | 28
  EOS, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  EOS, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 43 | 28
  EOS, pre-vacc. ABOVE, Month 7 ABOVE | 34 | 16
  EOS, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 19 | 10
  EOS, pre-vacc. BELOW, Month 7 NORMAL | 17 | 9
  EOS, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 19 | 10
  EOS, pre-vacc. BELOW, Month 7 BELOW | 2 | 1
  EOS, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 19 | 10
  EOS, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  EOS, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 155 | 67
  EOS, pre-vacc. NORMAL, Month 7 NORMAL | 134 | 56
  EOS, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 155 | 67
  EOS, pre-vacc. NORMAL, Month 7 BELOW | 3 | 2
  EOS, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 155 | 67
  EOS, pre-vacc. NORMAL, Month 7 ABOVE | 18 | 9
  HC, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 75 | 33
  HC, pre-vacc. BELOW, Month 7 NORMAL | 16 | 7
  HC, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 75 | 33
  HC, pre-vacc. BELOW, Month 7 BELOW | 59 | 26
  HC, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 75 | 33
  HC, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  HC, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 142 | 72
  HC, pre-vacc. NORMAL, Month 7 NORMAL | 104 | 52
  HC, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 142 | 72
  HC, pre-vacc. NORMAL, Month 7 BELOW | 38 | 20
  HC, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 142 | 72
  HC, pre-vacc. NORMAL, Month 7 ABOVE | 0 | 0
  LYM, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 77 | 41
  LYM, pre-vacc. ABOVE, Month 7 NORMAL | 23 | 11
  LYM, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 77 | 41
  LYM, pre-vacc. ABOVE, Month 7 BELOW | 4 | 3
  LYM, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 77 | 41
  LYM, pre-vacc. ABOVE, Month 7 ABOVE | 50 | 27
  LYM, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 41 | 19
  LYM, pre-vacc. BELOW, Month 7 NORMAL | 23 | 8
  LYM, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 41 | 19
  LYM, pre-vacc. BELOW, Month 7 BELOW | 11 | 6
  LYM, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 41 | 19
  LYM, pre-vacc. BELOW, Month 7 ABOVE | 7 | 5
  LYM, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 99 | 45
  LYM, pre-vacc. NORMAL, Month 7 NORMAL | 47 | 19
  LYM, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 99 | 45
  LYM, pre-vacc. NORMAL, Month 7 BELOW | 17 | 2
  LYM, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 99 | 45
  LYM, pre-vacc. NORMAL, Month 7 ABOVE | 35 | 24
  MON, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 48 | 35
  MON, pre-vacc. ABOVE, Month 7 NORMAL | 17 | 4
  MON, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 48 | 35
  MON, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  MON, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 48 | 35
  MON, pre-vacc. ABOVE, Month 7 ABOVE | 31 | 31
  MON, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 169 | 70
  MON, pre-vacc. NORMAL, Month 7 NORMAL | 108 | 45
  MON, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 169 | 70
  MON, pre-vacc. NORMAL, Month 7 BELOW | 0 | 0
  MON, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 169 | 70
  MON, pre-vacc. NORMAL, Month 7 ABOVE | 61 | 25
  NEU, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 8 | 3
  NEU, pre-vacc. ABOVE, Month 7 NORMAL | 0 | 0
  NEU, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 8 | 3
  NEU, pre-vacc. ABOVE, Month 7 BELOW | 7 | 3
  NEU, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 8 | 3
  NEU, pre-vacc. ABOVE, Month 7 ABOVE | 1 | 0
  NEU, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 176 | 91
  NEU, pre-vacc. BELOW, Month 7 NORMAL | 9 | 4
  NEU, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 176 | 91
  NEU, pre-vacc. BELOW, Month 7 BELOW | 165 | 86
  NEU, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 176 | 91
  NEU, pre-vacc. BELOW, Month 7 ABOVE | 2 | 1
  NEU, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 33 | 11
  NEU, pre-vacc. NORMAL, Month 7 NORMAL | 4 | 1
  NEU, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 33 | 11
  NEU, pre-vacc. NORMAL, Month 7 BELOW | 26 | 10
  NEU, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 33 | 11
  NEU, pre-vacc. NORMAL, Month 7 ABOVE | 3 | 0
  PLA, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 17 | 6
  PLA, pre-vacc. ABOVE, Month 7 NORMAL | 10 | 4
  PLA, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 17 | 6
  PLA, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  PLA, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 17 | 6
  PLA, pre-vacc. ABOVE, Month 7 ABOVE | 7 | 2
  PLA. pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 2 | 3
  PLA. pre-vacc. BELOW, Month 7 NORMAL | 1 | 0
  PLA. pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 2 | 3
  PLA. pre-vacc. BELOW, Month 7 BELOW | 1 | 2
  PLA. pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 2 | 3
  PLA. pre-vacc. BELOW, Month 7 ABOVE | 0 | 1
  PLA, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 198 | 96
  PLA, pre-vacc. NORMAL, Month 7 NORMAL | 194 | 96
  PLA, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 198 | 96
  PLA, pre-vacc. NORMAL, Month 7 BELOW | 0 | 0
  PLA, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 198 | 96
  PLA, pre-vacc. NORMAL, Month 7 ABOVE | 4 | 0
  RBC, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 29 | 11
  RBC, pre-vacc. BELOW, Month 7 NORMAL | 10 | 3
  RBC, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 29 | 11
  RBC, pre-vacc. BELOW, Month 7 BELOW | 19 | 8
  RBC, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 29 | 11
  RBC, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  RBC, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 188 | 94
  RBC, pre-vacc. NORMAL, Month 7 NORMAL | 176 | 89
  RBC, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 188 | 94
  RBC, pre-vacc. NORMAL, Month 7 BELOW | 12 | 5
  RBC, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 188 | 94
  RBC, pre-vacc. NORMAL, Month 7 ABOVE | 0 | 0
  WBC, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 9 | 7
  WBC, pre-vacc. ABOVE, Month 7 NORMAL | 6 | 6
  WBC, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 9 | 7
  WBC, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  WBC, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 9 | 7
  WBC, pre-vacc. ABOVE, Month 7 ABOVE | 3 | 1
  WBC, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 21 | 12
  WBC, pre-vacc. BELOW, Month 7 NORMAL | 5 | 6
  WBC, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 21 | 12
  WBC, pre-vacc. BELOW, Month 7 BELOW | 16 | 6
  WBC, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 21 | 12
  WBC, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  WBC, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 187 | 86
  WBC, pre-vacc. NORMAL, Month 7 NORMAL | 158 | 72
  WBC, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 187 | 86
  WBC, pre-vacc. NORMAL, Month 7 BELOW | 26 | 13
  WBC, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 187 | 86
  WBC, pre-vacc. NORMAL, Month 7 ABOVE | 3 | 1

12. Secondary Outcome: Number of Tanzanian Subjects With Clinically Relevant Abnormalities in Parameters Assessed
Description: as for outcome 11
Time Frame: At Month 7
Population: The analysis was performed on the Total Vaccinated cohort on Tanzanian subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 187 | 96
Participants
  ALT, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 3 | 3
  ALT, pre-vacc. ABOVE, Month 7 NORMAL | 2 | 2
  ALT, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 3 | 3
  ALT, pre-vacc. ABOVE, Month 7 BELOW | 0 | 1
  ALT, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 3 | 3
  ALT, pre-vacc. ABOVE, Month 7 ABOVE | 1 | 0
  ALT, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 13 | 11
  ALT, pre-vacc. BELOW, Month 7 NORMAL | 7 | 3
  ALT, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 13 | 11
  ALT, pre-vacc. BELOW, Month 7 BELOW | 6 | 8
  ALT, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 13 | 11
  ALT, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  ALT, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 183 | 85
  ALT, pre-vacc. NORMAL, Month 7 NORMAL | 144 | 65
  ALT, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 183 | 85
  ALT, pre-vacc. NORMAL, Month 7 BELOW | 39 | 20
  ALT, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 183 | 85
  ALT, pre-vacc. NORMAL, Month 7 ABOVE | 0 | 0
  BAS, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 21 | 12
  BAS, pre-vacc. ABOVE, Month 7 NORMAL | 19 | 12
  BAS, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 21 | 12
  BAS, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  BAS, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 21 | 12
  BAS, pre-vacc. ABOVE, Month 7 ABOVE | 2 | 0
  BAS, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 178 | 87
  BAS, pre-vacc. NORMAL, Month 7 NORMAL | 163 | 81
  BAS, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 178 | 87
  BAS, pre-vacc. NORMAL, Month 7 BELOW | 0 | 0
  BAS, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 178 | 87
  BAS, pre-vacc. NORMAL, Month 7 ABOVE | 15 | 6
  CREA, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 43 | 14
  CREA, pre-vacc. BELOW, Month 7 NORMAL | 2 | 2
  CREA, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 43 | 14
  CREA, pre-vacc. BELOW, Month 7 BELOW | 41 | 12
  CREA, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 43 | 14
  CREA, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  CREA, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 156 | 85
  CREA, pre-vacc. NORMAL, Month 7 NORMAL | 40 | 14
  CREA, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 156 | 85
  CREA, pre-vacc. NORMAL, Month 7 BELOW | 116 | 71
  CREA, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 156 | 85
  CREA, pre-vacc. NORMAL, Month 7 ABOVE | 0 | 0
  EOS, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 76 | 39
  EOS, pre-vacc. ABOVE, Month 7 NORMAL | 14 | 4
  EOS, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 76 | 39
  EOS, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  EOS, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 76 | 39
  EOS, pre-vacc. ABOVE, Month 7 ABOVE | 61 | 35
  EOS, pre-vacc. ABOVE, Month 7 MISSING: number analyzed (Participants) | 76 | 39
  EOS, pre-vacc. ABOVE, Month 7 MISSING | 1 | 0
  EOS, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 123 | 60
  EOS, pre-vacc. NORMAL, Month 7 NORMAL | 92 | 52
  EOS, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 123 | 60
  EOS, pre-vacc. NORMAL, Month 7 BELOW | 0 | 0
  EOS, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 123 | 60
  EOS, pre-vacc. NORMAL, Month 7 ABOVE | 31 | 8
  HC, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 1 | 0
  HC, pre-vacc. ABOVE, Month 7 NORMAL | 1 | 0
  HC, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 1 | 0
  HC, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  HC, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 1 | 0
  HC, pre-vacc. ABOVE, Month 7 ABOVE | 0 | 0
  HC, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 60 | 35
  HC, pre-vacc. BELOW, Month 7 NORMAL | 20 | 6
  HC, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 60 | 35
  HC, pre-vacc. BELOW, Month 7 BELOW | 40 | 29
  HC, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 60 | 35
  HC, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  HC, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 138 | 64
  HC, pre-vacc. NORMAL, Month 7 NORMAL | 118 | 51
  HC, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 138 | 64
  HC, pre-vacc. NORMAL, Month 7 BELOW | 20 | 13
  HC, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 138 | 64
  HC, pre-vacc. NORMAL, Month 7 ABOVE | 0 | 0
  LYM, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 20 | 8
  LYM, pre-vacc. ABOVE, Month 7 NORMAL | 12 | 7
  LYM, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 20 | 8
  LYM, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  LYM, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 20 | 8
  LYM, pre-vacc. ABOVE, Month 7 ABOVE | 8 | 1
  LYM, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 179 | 91
  LYM, pre-vacc. NORMAL, Month 7 NORMAL | 166 | 81
  LYM, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 179 | 91
  LYM, pre-vacc. NORMAL, Month 7 BELOW | 3 | 0
  LYM, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 179 | 91
  LYM, pre-vacc. NORMAL, Month 7 ABOVE | 10 | 10
  MON, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 12 | 7
  MON, pre-vacc. ABOVE, Month 7 NORMAL | 6 | 6
  MON, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 12 | 7
  MON, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  MON, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 12 | 7
  MON, pre-vacc. ABOVE, Month 7 ABOVE | 6 | 1
  MON, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 187 | 92
  MON, pre-vacc. NORMAL, Month 7 NORMAL | 180 | 85
  MON, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 187 | 92
  MON, pre-vacc. NORMAL, Month 7 BELOW | 0 | 0
  MON, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 187 | 92
  MON, pre-vacc. NORMAL, Month 7 ABOVE | 7 | 7
  NEU, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 36 | 16
  NEU, pre-vacc. BELOW, Month 7 NORMAL | 13 | 9
  NEU, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 36 | 16
  NEU, pre-vacc. BELOW, Month 7 BELOW | 22 | 7
  NEU, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 36 | 16
  NEU, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  NEU, pre-vacc. BELOW, Month 7 MISSING: number analyzed (Participants) | 36 | 16
  NEU, pre-vacc. BELOW, Month 7 MISSING | 1 | 0
  NEU, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 163 | 83
  NEU, pre-vacc. NORMAL, Month 7 NORMAL | 145 | 70
  NEU, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 163 | 83
  NEU, pre-vacc. NORMAL, Month 7 BELOW | 17 | 13
  NEU, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 163 | 83
  NEU, pre-vacc. NORMAL, Month 7 ABOVE | 1 | 0
  PLA, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 10 | 3
  PLA, pre-vacc. ABOVE, Month 7 NORMAL | 7 | 1
  PLA, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 10 | 3
  PLA, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  PLA, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 10 | 3
  PLA, pre-vacc. ABOVE, Month 7 ABOVE | 3 | 2
  PLA, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 5 | 0
  PLA, pre-vacc. BELOW, Month 7 NORMAL | 4 | 0
  PLA, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 5 | 0
  PLA, pre-vacc. BELOW, Month 7 BELOW | 1 | 0
  PLA, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 5 | 0
  PLA, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  PLA, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 184 | 96
  PLA, pre-vacc. NORMAL, Month 7 NORMAL | 180 | 92
  PLA, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 184 | 96
  PLA, pre-vacc. NORMAL, Month 7 BELOW | 2 | 0
  PLA, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 184 | 96
  PLA, pre-vacc. NORMAL, Month 7 ABOVE | 2 | 4
  RBC, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 11 | 7
  RBC, pre-vacc. ABOVE, Month 7 NORMAL | 6 | 4
  RBC, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 11 | 7
  RBC, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  RBC, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 11 | 7
  RBC, pre-vacc. ABOVE, Month 7 ABOVE | 5 | 3
  RBC, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 2 | 1
  RBC, pre-vacc. BELOW, Month 7 NORMAL | 1 | 0
  RBC, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 2 | 1
  RBC, pre-vacc. BELOW, Month 7 BELOW | 1 | 1
  RBC, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 2 | 1
  RBC, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  RBC, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 186 | 91
  RBC, pre-vacc. NORMAL, Month 7 NORMAL | 177 | 90
  RBC, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 186 | 91
  RBC, pre-vacc. NORMAL, Month 7 BELOW | 5 | 0
  RBC, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 186 | 91
  RBC, pre-vacc. NORMAL, Month 7 ABOVE | 4 | 1
  WBC, pre-vacc. ABOVE, Month 7 NORMAL: number analyzed (Participants) | 17 | 7
  WBC, pre-vacc. ABOVE, Month 7 NORMAL | 13 | 6
  WBC, pre-vacc. ABOVE, Month 7 BELOW: number analyzed (Participants) | 17 | 7
  WBC, pre-vacc. ABOVE, Month 7 BELOW | 0 | 0
  WBC, pre-vacc. ABOVE, Month 7 ABOVE: number analyzed (Participants) | 17 | 7
  WBC, pre-vacc. ABOVE, Month 7 ABOVE | 4 | 1
  WBC, pre-vacc. BELOW, Month 7 NORMAL: number analyzed (Participants) | 0 | 2
  WBC, pre-vacc. BELOW, Month 7 NORMAL | 0 | 2
  WBC, pre-vacc. BELOW, Month 7 BELOW: number analyzed (Participants) | 0 | 2
  WBC, pre-vacc. BELOW, Month 7 BELOW | 0 | 0
  WBC, pre-vacc. BELOW, Month 7 ABOVE: number analyzed (Participants) | 0 | 2
  WBC, pre-vacc. BELOW, Month 7 ABOVE | 0 | 0
  WBC, pre-vacc. NORMAL, Month 7 NORMAL: number analyzed (Participants) | 182 | 90
  WBC, pre-vacc. NORMAL, Month 7 NORMAL | 177 | 86
  WBC, pre-vacc. NORMAL, Month 7 BELOW: number analyzed (Participants) | 182 | 90
  WBC, pre-vacc. NORMAL, Month 7 BELOW | 4 | 2
  WBC, pre-vacc. NORMAL, Month 7 ABOVE: number analyzed (Participants) | 182 | 90
  WBC, pre-vacc. NORMAL, Month 7 ABOVE | 1 | 2

13. Secondary Outcome: Number of Senegalese Subjects With Clinically Relevant Abnormalities in Parameters Assessed
Description: as for outcome 11
Time Frame: At Month 12
Population: The analysis was performed on the Total Vaccinated cohort on Senegalese subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 211 | 102
Participants
  ALT, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 8 | 4
  ALT, pre-vacc. ABOVE, Month 12 NORMAL | 8 | 4
  ALT, pre-vacc.ABOVE, Month 12 BELOW: number analyzed (Participants) | 8 | 4
  ALT, pre-vacc.ABOVE, Month 12 BELOW | 0 | 0
  ALT, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 8 | 4
  ALT, pre-vacc. ABOVE, Month 12 ABOVE | 0 | 0
  ALT, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 38 | 17
  ALT, pre-vacc. BELOW, Month 12 NORMAL | 17 | 9
  ALT, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 38 | 17
  ALT, pre-vacc. BELOW, Month 12 BELOW | 21 | 8
  ALT, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 38 | 17
  ALT, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  ALT, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 165 | 81
  ALT, pre-vacc. NORMAL, Month 12 NORMAL | 139 | 61
  ALT, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 165 | 81
  ALT, pre-vacc. NORMAL, Month 12 BELOW | 24 | 17
  ALT, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 165 | 81
  ALT, pre-vacc. NORMAL, Month 12 ABOVE | 2 | 3
  BAS, pre-vacc. NORMAL, Month 12 NORMAL | 210 | 102
  BAS, pre-vacc. NORMAL, Month 12 BELOW | 0 | 0
  BAS, pre-vacc. NORMAL, Month 12 ABOVE | 1 | 0
  CREA, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 2 | 1
  CREA, pre-vacc. ABOVE, Month 12 NORMAL | 1 | 0
  CREA, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 2 | 1
  CREA, pre-vacc. ABOVE, Month 12 BELOW | 0 | 1
  CREA, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 2 | 1
  CREA, pre-vacc. ABOVE, Month 12 ABOVE | 1 | 0
  CREA, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 56 | 29
  CREA, pre-vacc. BELOW, Month 12 NORMAL | 13 | 6
  CREA, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 56 | 29
  CREA, pre-vacc. BELOW, Month 12 BELOW | 43 | 23
  CREA, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 56 | 29
  CREA, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  CREA, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 153 | 72
  CREA, pre-vacc. NORMAL, Month 12 NORMAL | 130 | 64
  CREA, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 153 | 72
  CREA, pre-vacc. NORMAL, Month 12 BELOW | 23 | 8
  CREA, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 153 | 72
  CREA, pre-vacc. NORMAL, Month 12 ABOVE | 0 | 0
  EOS, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 43 | 28
  EOS, pre-vacc. ABOVE, Month 12 NORMAL | 14 | 11
  EOS, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 43 | 28
  EOS, pre-vacc. ABOVE, Month 12 BELOW | 1 | 0
  EOS, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 43 | 28
  EOS, pre-vacc. ABOVE, Month 12 ABOVE | 28 | 17
  EOS, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 19 | 10
  EOS, pre-vacc. BELOW, Month 12 NORMAL | 13 | 6
  EOS, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 19 | 10
  EOS, pre-vacc. BELOW, Month 12 BELOW | 6 | 3
  EOS, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 19 | 10
  EOS, pre-vacc. BELOW, Month 12 ABOVE | 0 | 1
  EOS, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 149 | 64
  EOS, pre-vacc. NORMAL, Month 12 NORMAL | 126 | 52
  EOS, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 149 | 64
  EOS, pre-vacc. NORMAL, Month 12 BELOW | 6 | 2
  EOS, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 149 | 64
  EOS, pre-vacc. NORMAL, Month 12 ABOVE | 17 | 10
  HC, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 71 | 33
  HC, pre-vacc. BELOW, Month 12 NORMAL | 15 | 10
  HC, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 71 | 33
  HC, pre-vacc. BELOW, Month 12 BELOW | 56 | 23
  HC, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 71 | 33
  HC, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  HC, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 140 | 69
  HC, pre-vacc. NORMAL, Month 12 NORMAL | 108 | 45
  HC, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 140 | 69
  HC, pre-vacc. NORMAL, Month 12 BELOW | 32 | 24
  HC, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 140 | 69
  HC, pre-vacc. NORMAL, Month 12 ABOVE | 0 | 0
  LYM, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 75 | 41
  LYM, pre-vacc. ABOVE, Month 12 NORMAL | 24 | 16
  LYM, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 75 | 41
  LYM, pre-vacc. ABOVE, Month 12 BELOW | 4 | 3
  LYM, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 75 | 41
  LYM, pre-vacc. ABOVE, Month 12 ABOVE | 47 | 22
  LYM, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 38 | 19
  LYM, pre-vacc. BELOW, Month 12 NORMAL | 9 | 8
  LYM, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 38 | 19
  LYM, pre-vacc. BELOW, Month 12 BELOW | 15 | 5
  LYM, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 38 | 19
  LYM, pre-vacc. BELOW, Month 12 ABOVE | 14 | 6
  LYM, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 98 | 42
  LYM, pre-vacc. NORMAL, Month 12 NORMAL | 48 | 24
  LYM, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 98 | 42
  LYM, pre-vacc. NORMAL, Month 12 BELOW | 27 | 4
  LYM, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 98 | 42
  LYM, pre-vacc. NORMAL, Month 12 ABOVE | 23 | 14
  MON, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 45 | 34
  MON, pre-vacc. ABOVE, Month 12 NORMAL | 13 | 10
  MON, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 45 | 34
  MON, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  MON, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 45 | 34
  MON, pre-vacc. ABOVE, Month 12 ABOVE | 32 | 24
  MON, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 166 | 68
  MON, pre-vacc. NORMAL, Month 12 NORMAL | 102 | 38
  MON, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 166 | 68
  MON, pre-vacc. NORMAL, Month 12 BELOW | 0 | 0
  MON, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 166 | 68
  MON, pre-vacc. NORMAL, Month 12 ABOVE | 64 | 30
  NEU, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 8 | 3
  NEU, pre-vacc. ABOVE, Month 12 NORMAL | 4 | 0
  NEU, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 8 | 3
  NEU, pre-vacc. ABOVE, Month 12 BELOW | 4 | 3
  NEU, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 8 | 3
  NEU, pre-vacc. ABOVE, Month 12 ABOVE | 0 | 0
  NEU, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 173 | 88
  NEU, pre-vacc. BELOW, Month 12 NORMAL | 11 | 5
  NEU, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 173 | 88
  NEU, pre-vacc. BELOW, Month 12 BELOW | 160 | 83
  NEU, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 173 | 88
  NEU, pre-vacc. BELOW, Month 12 ABOVE | 2 | 0
  NEU, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 30 | 11
  NEU, pre-vacc. NORMAL, Month 12 NORMAL | 7 | 1
  NEU, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 30 | 11
  NEU, pre-vacc. NORMAL, Month 12 BELOW | 22 | 9
  NEU, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 30 | 11
  NEU, pre-vacc. NORMAL, Month 12 ABOVE | 1 | 1
  PLA, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 17 | 6
  PLA, pre-vacc. ABOVE, Month 12 NORMAL | 13 | 4
  PLA, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 17 | 6
  PLA, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  PLA, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 17 | 6
  PLA, pre-vacc. ABOVE, Month 12 ABOVE | 4 | 2
  PLA. pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 2 | 3
  PLA. pre-vacc. BELOW, Month 12 NORMAL | 1 | 1
  PLA. pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 2 | 3
  PLA. pre-vacc. BELOW, Month 12 BELOW | 1 | 2
  PLA. pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 2 | 3
  PLA. pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  PLA, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 192 | 93
  PLA, pre-vacc. NORMAL, Month 12 NORMAL | 188 | 93
  PLA, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 198 | 93
  PLA, pre-vacc. NORMAL, Month 12 BELOW | 3 | 0
  PLA, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 198 | 93
  PLA, pre-vacc. NORMAL, Month 12 ABOVE | 1 | 0
  RBC, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 27 | 11
  RBC, pre-vacc. BELOW, Month 12 NORMAL | 8 | 5
  RBC, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 27 | 11
  RBC, pre-vacc. BELOW, Month 12 BELOW | 19 | 6
  RBC, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 27 | 11
  RBC, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  RBC, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 184 | 91
  RBC, pre-vacc. NORMAL, Month 12 NORMAL | 169 | 80
  RBC, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 184 | 91
  RBC, pre-vacc. NORMAL, Month 12 BELOW | 15 | 11
  RBC, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 184 | 91
  RBC, pre-vacc. NORMAL, Month 12 ABOVE | 0 | 0
  WBC, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 8 | 7
  WBC, pre-vacc. ABOVE, Month 12 NORMAL | 6 | 7
  WBC, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 8 | 7
  WBC, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  WBC, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 8 | 7
  WBC, pre-vacc. ABOVE, Month 12 ABOVE | 2 | 0
  WBC, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 19 | 12
  WBC, pre-vacc. BELOW, Month 12 NORMAL | 10 | 5
  WBC, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 19 | 12
  WBC, pre-vacc. BELOW, Month 12 BELOW | 9 | 7
  WBC, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 19 | 12
  WBC, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  WBC, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 184 | 83
  WBC, pre-vacc. NORMAL, Month 12 NORMAL | 156 | 64
  WBC, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 184 | 83
  WBC, pre-vacc. NORMAL, Month 12 BELOW | 22 | 16
  WBC, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 184 | 83
  WBC, pre-vacc. NORMAL, Month 12 ABOVE | 6 | 3

14. Secondary Outcome: Number of Tanzanian Subjects With Clinically Relevant Abnormalities in Parameters Assessed
Description: as for outcome 11
Time Frame: At Month 12
Population: The analysis was performed on the Total Vaccinated cohort on Tanzanian subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 194 | 100
Participants
  ALT, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 3 | 4
  ALT, pre-vacc. ABOVE, Month 12 NORMAL | 2 | 2
  ALT, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 3 | 4
  ALT, pre-vacc. ABOVE, Month 12 BELOW | 0 | 1
  ALT, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 3 | 4
  ALT, pre-vacc. ABOVE, Month 12 ABOVE | 1 | 1
  ALT, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 13 | 11
  ALT, pre-vacc. BELOW, Month 12 NORMAL | 12 | 8
  ALT, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 13 | 11
  ALT, pre-vacc. BELOW, Month 12 BELOW | 1 | 3
  ALT, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 13 | 11
  ALT, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  ALT, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 190 | 87
  ALT, pre-vacc. NORMAL, Month 12 NORMAL | 166 | 73
  ALT, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 190 | 87
  ALT, pre-vacc. NORMAL, Month 12 BELOW | 24 | 13
  ALT, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 190 | 87
  ALT, pre-vacc. NORMAL, Month 12 ABOVE | 0 | 1
  BAS, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 23 | 13
  BAS, pre-vacc. ABOVE, Month 12 NORMAL | 21 | 12
  BAS, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 23 | 13
  BAS, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  BAS, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 23 | 13
  BAS, pre-vacc. ABOVE, Month 12 ABOVE | 2 | 1
  BAS, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 183 | 89
  BAS, pre-vacc. NORMAL, Month 12 NORMAL | 174 | 81
  BAS, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 183 | 89
  BAS, pre-vacc. NORMAL, Month 12 BELOW | 0 | 0
  BAS, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 183 | 89
  BAS, pre-vacc. NORMAL, Month 12 ABOVE | 9 | 8
  CREA, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 42 | 14
  CREA, pre-vacc. BELOW, Month 12 NORMAL | 2 | 0
  CREA, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 42 | 14
  CREA, pre-vacc. BELOW, Month 12 BELOW | 40 | 14
  CREA, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 42 | 14
  CREA, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  CREA, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 164 | 88
  CREA, pre-vacc. NORMAL, Month 12 NORMAL | 48 | 19
  CREA, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 164 | 88
  CREA, pre-vacc. NORMAL, Month 12 BELOW | 116 | 69
  CREA, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 164 | 88
  CREA, pre-vacc. NORMAL, Month 12 ABOVE | 0 | 0
  EOS, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 79 | 43
  EOS, pre-vacc. ABOVE, Month 12 NORMAL | 22 | 10
  EOS, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 79 | 43
  EOS, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  EOS, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 79 | 43
  EOS, pre-vacc. ABOVE, Month 12 ABOVE | 57 | 33
  EOS, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 127 | 59
  EOS, pre-vacc. NORMAL, Month 12 NORMAL | 93 | 48
  EOS, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 127 | 59
  EOS, pre-vacc. NORMAL, Month 12 BELOW | 0 | 0
  EOS, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 127 | 59
  EOS, pre-vacc. NORMAL, Month 12 ABOVE | 34 | 11
  HC, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 63 | 38
  HC, pre-vacc. BELOW, Month 12 NORMAL | 29 | 10
  HC, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 63 | 38
  HC, pre-vacc. BELOW, Month 12 BELOW | 34 | 28
  HC, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 63 | 38
  HC, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  HC, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 143 | 64
  HC, pre-vacc. NORMAL, Month 12 NORMAL | 107 | 48
  HC, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 143 | 64
  HC, pre-vacc. NORMAL, Month 12 BELOW | 36 | 16
  HC, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 143 | 64
  HC, pre-vacc. NORMAL, Month 12 ABOVE | 0 | 0
  LYM, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 18 | 8
  LYM, pre-vacc. ABOVE, Month 12 NORMAL | 9 | 3
  LYM, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 18 | 8
  LYM, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  LYM, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 18 | 8
  LYM, pre-vacc. ABOVE, Month 12 ABOVE | 9 | 5
  LYM, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 188 | 94
  LYM, pre-vacc. NORMAL, Month 12 NORMAL | 168 | 81
  LYM, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 188 | 94
  LYM, pre-vacc. NORMAL, Month 12 BELOW | 0 | 2
  LYM, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 188 | 94
  LYM, pre-vacc. NORMAL, Month 12 ABOVE | 20 | 11
  MON, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 12 | 7
  MON, pre-vacc. ABOVE, Month 12 NORMAL | 8 | 6
  MON, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 12 | 7
  MON, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  MON, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 12 | 7
  MON, pre-vacc. ABOVE, Month 12 ABOVE | 4 | 1
  MON, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 194 | 95
  MON, pre-vacc. NORMAL, Month 12 NORMAL | 184 | 88
  MON, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 194 | 95
  MON, pre-vacc. NORMAL, Month 12 BELOW | 0 | 0
  MON, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 194 | 95
  MON, pre-vacc. NORMAL, Month 12 ABOVE | 10 | 7
  NEU, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 36 | 17
  NEU, pre-vacc. BELOW, Month 12 NORMAL | 18 | 6
  NEU, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 36 | 17
  NEU, pre-vacc. BELOW, Month 12 BELOW | 18 | 11
  NEU, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 36 | 17
  NEU, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  NEU, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 170 | 85
  NEU, pre-vacc. NORMAL, Month 12 NORMAL | 138 | 72
  NEU, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 170 | 85
  NEU, pre-vacc. NORMAL, Month 12 BELOW | 32 | 13
  NEU, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 170 | 85
  NEU, pre-vacc. NORMAL, Month 12 ABOVE | 0 | 0
  PLA, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 10 | 2
  PLA, pre-vacc. ABOVE, Month 12 NORMAL | 8 | 1
  PLA, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 10 | 2
  PLA, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  PLA, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 10 | 2
  PLA, pre-vacc. ABOVE, Month 12 ABOVE | 2 | 1
  PLA, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 5 | 0
  PLA, pre-vacc. BELOW, Month 12 NORMAL | 5 | 0
  PLA, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 5 | 0
  PLA, pre-vacc. BELOW, Month 12 BELOW | 0 | 0
  PLA, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 5 | 0
  PLA, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  PLA, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 191 | 100
  PLA, pre-vacc. NORMAL, Month 12 NORMAL | 185 | 96
  PLA, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 191 | 100
  PLA, pre-vacc. NORMAL, Month 12 BELOW | 1 | 2
  PLA, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 191 | 100
  PLA, pre-vacc. NORMAL, Month 12 ABOVE | 5 | 2
  RBC, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 10 | 7
  RBC, pre-vacc. ABOVE, Month 12 NORMAL | 5 | 3
  RBC, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 10 | 7
  RBC, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  RBC, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 10 | 7
  RBC, pre-vacc. ABOVE, Month 12 ABOVE | 5 | 4
  RBC, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 3 | 2
  RBC, pre-vacc. BELOW, Month 12 NORMAL | 2 | 0
  RBC, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 3 | 2
  RBC, pre-vacc. BELOW, Month 12 BELOW | 1 | 2
  RBC, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 3 | 2
  RBC, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  RBC, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 193 | 93
  RBC, pre-vacc. NORMAL, Month 12 NORMAL | 182 | 91
  RBC, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 193 | 93
  RBC, pre-vacc. NORMAL, Month 12 BELOW | 6 | 2
  RBC, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 193 | 93
  RBC, pre-vacc. NORMAL, Month 12 ABOVE | 5 | 0
  WBC, pre-vacc. ABOVE, Month 12 NORMAL: number analyzed (Participants) | 17 | 6
  WBC, pre-vacc. ABOVE, Month 12 NORMAL | 12 | 5
  WBC, pre-vacc. ABOVE, Month 12 BELOW: number analyzed (Participants) | 17 | 6
  WBC, pre-vacc. ABOVE, Month 12 BELOW | 0 | 0
  WBC, pre-vacc. ABOVE, Month 12 ABOVE: number analyzed (Participants) | 17 | 6
  WBC, pre-vacc. ABOVE, Month 12 ABOVE | 5 | 1
  WBC, pre-vacc. BELOW, Month 12 NORMAL: number analyzed (Participants) | 0 | 2
  WBC, pre-vacc. BELOW, Month 12 NORMAL | 0 | 2
  WBC, pre-vacc. BELOW, Month 12 BELOW: number analyzed (Participants) | 0 | 2
  WBC, pre-vacc. BELOW, Month 12 BELOW | 0 | 0
  WBC, pre-vacc. BELOW, Month 12 ABOVE: number analyzed (Participants) | 0 | 2
  WBC, pre-vacc. BELOW, Month 12 ABOVE | 0 | 0
  WBC, pre-vacc. NORMAL, Month 12 NORMAL: number analyzed (Participants) | 189 | 94
  WBC, pre-vacc. NORMAL, Month 12 NORMAL | 165 | 85
  WBC, pre-vacc. NORMAL, Month 12 BELOW: number analyzed (Participants) | 189 | 94
  WBC, pre-vacc. NORMAL, Month 12 BELOW | 14 | 5
  WBC, pre-vacc. NORMAL, Month 12 ABOVE: number analyzed (Participants) | 189 | 94
  WBC, pre-vacc. NORMAL, Month 12 ABOVE | 10 | 4

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: within 7 days (Day 0-6) after vaccination; Unsolicited AEs: within 30 days (Day 0-29) after any vaccination; SAEs: during the whole study period (from Day 0 up to Month 12).
Arm/Group | Cervarix Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/450 | 0/226
Serious Adverse Events (participants affected / at risk) | 17/450 | 14/226
Other Adverse Events (participants affected / at risk) | 433/450 | 216/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=450) | Placebo Group (N=226)
Malaria (Infections and infestations) | 10 | 11
Urinary tract infection (Infections and infestations) | 0 | 3
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Burn infection (Infections and infestations) | 0 | 1
Dysentery (Infections and infestations) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Neuropathy vitamin b6 deficiency (Nervous system disorders) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pyomyositis (Infections and infestations) | 1 | 0
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=450) | Placebo Group (N=226)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 16 (17) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Adenoiditis (Infections and infestations) | 1 (1) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Amoebiasis (Infections and infestations) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 79 (97) | 36 (41)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Body tinea (Infections and infestations) | 7 (7) | 3 (3)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 5 (5) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 8 (8) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 7 (8)
Cutaneous larva migrans (Infections and infestations) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 6 (6) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 23 (25) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 5 (5) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye allergy (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 4 (4) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 111 (130) | 42 (50)
Fungal infection (Infections and infestations) | 2 (2) | 1 (1)
Fungal skin infection (Infections and infestations) | 4 (4) | 2 (2)
Gastritis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 118 (143) | 56 (66)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Genital discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 201 (298) | 116 (157)
Helminthic infection (Infections and infestations) | 8 (8) | 1 (1)
Hookworm infection (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 8 (8) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 56 (66) | 38 (44)
Measles (Infections and infestations) | 0 (0) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 90 (113) | 38 (46)
Myopia (Eye disorders) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (10) | 12 (12)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (6)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 376 (779) | 168 (279)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 4 (5) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 147 (235) | 71 (110)
Rash (Skin and subcutaneous tissue disorders) | 71 (84) | 33 (38)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Swelling (General disorders) | 74 (86) | 27 (32)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 4 (4) | 2 (2)
Toothache (Gastrointestinal disorders) | 6 (6) | 3 (3)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trichuriasis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 68 (81) | 28 (33)
Vaginal discharge (Reproductive system and breast disorders) | 6 (6) | 4 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 13 (15) | 3 (4)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vulvitis (Infections and infestations) | 1 (1) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.